CLINICAL TRIAL: NCT04504812
Title: A Sequenced Strategy for Improving Outcomes in People With Knee Osteoarthritis Pain
Acronym: SKOAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00238678; 1UG3AR077360-01 (NIH)
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Knee Osteoarthritis
Keywords: osteoarthritis; duloxetine; painTRAINER; hyaluronic acid injection; genicular nerve block; radiofrequency ablation
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Duloxetine Hydrochloride; Injections, Intra-Articular; Practice Guidelines as Topic

STUDY DESIGN:
Intervention Model Description: Using a stepped care model, Phase 1 participants will be randomly assigned to minimally invasive treatments, including best practices, best practices plus duloxetine, and best practices plus duloxetine combined with a web-based pain coping skills training program. Those who note interest in additional treatment following completion of Phase 1, as well as those that are not eligible for Phase 1 treatment, will be randomly assigned to more aggressive procedures: intra-articular hyaluronic acid, steroid and local anesthetic injection, or a nerve procedure that would either include a long acting block or nerve ablation. Interim analyses will be completed for both phases, and pre-specified stopping rules will determine if all study arms will continue. Modified Intention to Treat (mITT) and per protocol analyses will be conducted.
Who Masked: Participant
Masking Description: Individuals randomized to a nerve procedure will be blinded to whether they have a long acting block or nerve ablation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Phase 1: Best Practices + Duloxetine (Active Comparator): Participants will receive Duloxetine and a prescription for guideline-recommended treatments for knee osteoarthritis, i.e., Best Practices. Best Practices can include topical or oral nonsteroidal anti-inflammatory drugs (NSAIDs), acetaminophen; physical therapy that may include aquatherapy; integrative treatments such as acupuncture, yoga, or a structured exercise program; and other non-invasive treatments.
  Phase 1 ended enrollment on April 12, 2024.
  Interventions: Drug: Duloxetine; Other: Best Practices
- Phase 1: Best Practices + Duloxetine + Pain coping skills (Active Comparator): Participants will receive Duloxetine, pain coping skills training, and a prescription for guideline-recommended treatments for knee osteoarthritis, i.e., Best Practices. Best Practices can include topical or oral nonsteroidal anti-inflammatory drugs (NSAIDs), acetaminophen; physical therapy that may include aquatherapy; integrative treatments such as acupuncture, yoga, or a structured exercise program; and other non-invasive treatments.
  Phase 1 ended enrollment on April 12, 2024.
  Interventions: Drug: Duloxetine; Behavioral: Pain Coping Skills Training; Other: Best Practices
- Phase 2: Intra-Articular Injection (HA+) (Active Comparator): Participants will receive an intra-articular injection of hyaluronic acid mixed with steroid and bupivacaine.
  Phase 2 ended enrollment on October 24, 2024.
  Interventions: Combination Product: Intra-Articular Injection
- Phase 2: Nerve Procedure: Long Acting Blocks (Active Comparator): Participants will receive a nerve blocking procedure, long-acting local anesthetic, and steroid injection.
  Phase 2 ended enrollment on October 24, 2024.
  Interventions: Procedure: Nerve Procedure with long acting blocks
- Phase 2: Nerve Procedure: Nerve Ablation (Active Comparator): Participants will receive a nerve ablation procedure and steroid injection.
  Phase 2 ended enrollment on October 24, 2024.
  Interventions: Procedure: Nerve Procedure with nerve ablation
- Phase 1: Best Practices (Active Comparator): Participants will receive a prescription for guideline-recommended treatments for knee osteoarthritis, i.e., Best Practices. Best Practices can include topical or oral nonsteroidal anti-inflammatory drugs (NSAIDs), acetaminophen; physical therapy that may include aquatherapy; integrative treatments such as acupuncture, yoga, or a structured exercise program; and other non-invasive treatments.
  Based on the pre-specified stopping rules described in Protocol section 13.2, the DSMB advised ceasing enrollment into Arm 1A (Best Practices). This recommendation was accepted by the sponsor and study investigators. Arm 1A (Best Practices) was closed on 11/29/2023.
  Interventions: Other: Best Practices

INTERVENTIONS:
Drug: Duloxetine — Duloxetine is a drug that is used to improve pain and function in people with knee osteoarthritis (KOA). Duloxetine is approved by the Food and Drug Administration (FDA) for the treatment of depression, anxiety disorder, fibromyalgia, and joint pain. It will be titrated up from 20 or 30mg according to a schedule provided by a study provider.
  Other Names: Cymbalta
  Arms: Phase 1: Best Practices + Duloxetine; Phase 1: Best Practices + Duloxetine + Pain coping skills
Combination Product: Intra-Articular Injection — Intra-Articular Injection is an injection of 3-6 milliliter (mL) hyaluronic acid (HA) mixed with 1 milliliter (mL) depo methylprednisolone (a steroid) and 2 mL 0.5% bupivacaine (an anesthetic) into the knee.
  Arms: Phase 2: Intra-Articular Injection (HA+)
Procedure: Nerve Procedure with long acting blocks — People assigned to receive this will have 1 milliliter (mL) of a long-acting local anesthetic (a.k.a. liposomal bupivacaine or EXPAREL) and steroid injected into the knee.
  Arms: Phase 2: Nerve Procedure: Long Acting Blocks
Procedure: Nerve Procedure with nerve ablation — People assigned to receive this will have heat applied to destroy the nerve signaling pain in the knee. Steroid will be administered after the procedure to reduce the risk of neuritis.
  Arms: Phase 2: Nerve Procedure: Nerve Ablation
Behavioral: Pain Coping Skills Training — Participants will be provided with a written manual that includes login information for the pain coping skills training website. The participants will be expected to log into the system weekly, work through the modules, and participate in skills practice. This intervention will be conducted in combination with best practices and duloxetine.
  Arms: Phase 1: Best Practices + Duloxetine + Pain coping skills
Other: Best Practices — Best Practices can include topical or oral nonsteroidal anti-inflammatory drugs (NSAIDs), acetaminophen; physical therapy that may include aquatherapy; integrative treatments such as acupuncture, yoga, or a structured exercise program; and other non-invasive treatments.
  Arms: Phase 1: Best Practices; Phase 1: Best Practices + Duloxetine; Phase 1: Best Practices + Duloxetine + Pain coping skills

SUMMARY:
There is an urgent public health need to reduce reliance on opioids for effective long-term pain management, particularly in knee osteoarthritis (KOA). This effectiveness trial will compare commonly recommended treatments to reduce pain and functional limitations in KOA.These results will lead to improved patient selection for treatment and inform evidence based guidelines by offering well-tested, effective, non-surgical alternatives.

DETAILED DESCRIPTION:
Knee osteoarthritis (KOA) is one of the leading causes of chronic pain and disability worldwide, affecting over 30% of older adults. It represents a major global health and economic burden to individuals and society. The rates of KOA have more than doubled in the past 70 years and continue to grow sharply, given increases in life expectancy and population body mass index (BMI). Surgery is often employed to treat KOA, but it is associated with a high rate of persistent pain, and is not a permanent solution. Numerous nonsurgical therapies have been advocated to treat pain in patients with KOA yet are not often used in clinical care. The limited pain relief and functional improvement seen in a subset of knee OA sufferers has led to a high rate of opioid use and disability in this population. The overarching goal of this study is to conduct a sequential parallel group randomized controlled trial (RCT) to evaluate the comparative effectiveness of conservative behavioral and non-opioid pharmacological treatments (Phase 1) and, among those that indicate interest in obtaining further treatment and those not eligible for conservative treatment, the benefits of procedural interventions (Phase 2). This study will also evaluate whether clinical and psychosocial phenotypes predict short- and longer-term treatment response. The results of this study will examine the effectiveness of each tested intervention and provide meaningful information regarding effectiveness across key subgroups of participants.

ELIGIBILITY:
Inclusion Criteria:

* Knee pain score of ≥4 and ≤ 9 on the Modified 4-Item BPI Pain Scale at pre-intervention screening
* Meets at least 1 of the 3 American College of Rheumatology (ACR) Classification criteria for knee osteoarthritis.

ACR criteria are:

1. At least three of the following using history and physical examination: age >50 years old; morning stiffness <30 minutes; crepitus on knee motion; bony tenderness; bony enlargement; no palpable warmth
2. At least one of the following using history, physical examination, and radiographic findings + the presence of osteophytes: age >50 years old; morning stiffness <30 minutes; crepitus on active motion and osteophytes
3. At least 5 of the following using history, physical examination, and laboratory findings: age >50 years old; morning stiffness <30 minutes; crepitus on knee motion; bony tenderness; bony enlargement; no palpable warmth; erythrocyte sedimentation rate (ESR) <40 mm/hour; Rheumatoid Factor (RF) <1:40; synovial fluid signs of osteoarthritis

Exclusion Criteria:

* <18 years of age
* Any inability to complete study procedures, including, but not limited to inadequate resources to mitigate low English language literacy
* Refusal of randomization
* Knee pain exclusions: Pain during an average of < 4 days per week over the past 3 months; pain in the index knee from a joint disease other than OA (e.g., infectious arthritis, rheumatoid arthritis, spondyloarthropathy)
* Medication exclusions: Report changes in analgesic medication dose within 2 weeks of baseline; oral morphine equivalent dose of > 90 mg/d at baseline
* Medical condition exclusions: Severe vision or hearing impairment or any signs of cognitive impairment that would prevent comprehension of consent procedures, study measures, or procedures; unstable medical condition that presents an absolute or relative contraindication for participation in both arms (e.g., unstable angina, congestive heart failure); poorly controlled serious psychiatric condition that could prevent full participation or affect outcomes (e.g., suicidal ideation, active psychosis, poorly controlled depression, active substance abuse [excluding tobacco, caffeine or moderate alcohol use])
* Knee-specific medical condition exclusions: History of bilateral knee joint replacement arthroplasty total knee arthroplasty (TKA) or TKA in the affected knee; partial replacements may be eligible depending on physician judgment; scheduled joint replacement; history of unilateral TKA and complaints of KOA pain limited to the operated knee; Intra-articular viscosupplementation, steroid injection or arthroscopic surgery in the index knee within 12 weeks of baseline
* Pregnancy by self-report, report of intention to become pregnant (Phase 1), or as determined by urine pregnancy screening (if Standard of Care at site) (Phase 2). Due to the unknown effects of duloxetine on the developing fetus and newborn, and the potential harms of fluoroscopy in pregnancy, women who are pregnant or lactating or intend to get pregnant will not be included in this study. Those of childbearing potential will be asked to use reliable contraception during the course of their participation in the study and to notify the study team if they become pregnant during participation. Definition of reliable birth control will be defined as: Female and male sterilization (female tubal ligation or occlusion, male vasectomy); long-acting reversible contraceptives (LARC) methods (intrauterine devices, hormonal implants); short-acting hormonal methods (pill, mini pills, patch, shot, vaginal ring); barrier methods (condoms, diaphragms, sponge, cervical cap)

Phase 1 specific Exclusion Criteria- An individual who meets any of the following criteria will be excluded from participation in Phase 1 of this study and will be enrolled and randomized directly into Phase 2:

* Known allergic reaction or medical condition that renders an individual unsuitable for Phase 1 study interventions, including closed-angle glaucoma, kidney disease (creatinine clearance < 30 mL/ min), severe liver disease, known adverse reaction to duloxetine or another selective serotonin-norepinephrine reuptake inhibitor (SNRI), bipolar disorder or mania, high likelihood of drug interactions that could lead to side effects (e.g., serotonin syndrome in people on multiple drugs that inhibit serotonin reuptake including monoamine oxidase (MAO) inhibitors).
* Report failed trial of an adequate dose of duloxetine to relieve KOA symptoms over a 1-month period
* Have tried and failed two of the following: NSAIDS, physical therapy (there are many physical therapies so clinicians should exercise their judgment as to what constitutes 'failed' therapy), or weight loss (need determined by clinician) and refuses participation in Phase 1
* End-stage renal disease
* Unreliable access to the internet on a daily basis, i.e., sufficient access to participate in the study and may include public library access, cafe/coffee shop spaces, access to a friend or neighbor's wifi or hotspot, etc. (reliability determined on a site-by-site basis)

Phase 2 specific exclusion criteria- An individual who meets any of the following is excluded from sequential participation in Phase 1 and then Phase 2, and will instead be randomized as a "solo" recruit into Phase 1:

* Inability to pay for interventions (insurance or otherwise)
* Medical condition exclusions: Untreated coagulopathy that could interfere with Phase 2 interventions; for automated implantable cardioverter-defibrillator that cannot be disabled before radiofrequency ablation (RFA), the investigator can consult cardiology, bioengineering or the device manufacturer before enrolling in phase 2 (i.e. not a definite exclusion criterion)
* Knee specific medical condition exclusions: Current local infection in the knee; ulcers or an open wound in the region of the index knee; underwent an adequate trial of any Phase 2 procedural study intervention in the study knee; severe needle phobia that cannot be addressed pharmacologically

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1937 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity as assessed by the Modified 4-item Brief Pain Inventory (BPI) Pain Scale | Change from Baseline to 8 weeks post-randomization (mITT) and to 8 weeks post-treatment (per protocol) in Phase 1; Change from Baseline to 12 weeks post-randomization (mITT) and to 12 weeks post-treatment (per protocol) in Phase 2
  The Modified 4-item BPI Pain scale consists of 3 items from BPI Pain Intensity and 1 item from BPI Pain Interference. This is a continuous measure that will be calculated as the average of worst, average, current knee pain, and pain upon walking. Change from baseline (BL) will be used in mITT analyses, and change from treatment will be used in per protocol analyses.

SECONDARY OUTCOMES:
Change in Pain Interference as assessed by the BPI | Change from Baseline to 8 weeks post-randomization (mITT) and to 8 weeks post-treatment (per protocol) in Phase 1; Change from Baseline to 12 weeks post-randomization (mITT) and to 12 weeks post-treatment (per protocol) in Phase 2
  The BPI Pain Interference domain assesses self-reported consequences of pain on relevant aspects of one's life. The BPI measures how much pain has interfered with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others, and sleep. BPI pain interference is typically scored as the mean of the seven interference items. BPI Interference ranges from 0-10 with higher scores reflecting greater pain interference in activities of daily living.
Change in Physical Functioning as assessed by the Knee Injury and Osteoarthritis Outcome Score (KOOS) | Change from baseline to 8 weeks post-randomization (mITT) and to 8 weeks post-treatment (per protocol) in Phase 1; Change from Baseline to 12 weeks post-randomization (mITT) and to 12 weeks post-treatment (per protocol) in Phase 2
  The KOOS evaluates function for participants with osteoarthritis of the knee that is related to injury and degeneration. The KOOS short form includes 12 items and measures pain, functional limitation and quality of life. Physical functioning questions cover everyday activities such as rising from sitting, standing getting in and out of the car and twisting/pivoting on the knee. Scores range from 0-100 with lower scores indicating worse knee symptoms.
Patient Global impression of Change (PGIC) | 8 weeks post-randomization (mITT) and 8 weeks post-treatment (per protocol) in Phase 1; 12 weeks post-randomization (mITT) and 12 weeks post-treatment (per protocol) in Phase 2
  The PGIC scale evaluates all aspects of participants' health and assesses if there has been an improvement or decline in clinical status. It is a 7-item scale that ranges between "a great deal worse" to "a great deal better." Higher scores reflect greater improvement in clinical status.
Change in Pain Intensity as assessed by the BPI | Change from baseline to 8 weeks post-randomization (mITT) and to 8 weeks post-treatment (per protocol) in Phase 1; Change from baseline to 12 weeks post-randomization (mITT) and to 12 weeks post-treatment (per protocol) in Phase 2
  The BPI Pain Interference domain assesses self-reported consequences of pain on relevant aspects of one's life. The BPI measures how much pain has interfered with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others, and sleep. BPI pain interference is typically scored as the mean of the seven interference items. BPI Interference ranges from 0-10 with higher scores reflecting greater pain interference in activities of daily living.
Compare Morphine Milligram Equivalent (MME) doses | Change from baseline to 8 weeks post-randomization (mITT) and to 8 weeks post-treatment (per protocol) in Phase 1; Change from baseline to 12 weeks post-randomization (mITT) and to 12 weeks post-treatment (per protocol) in Phase 2
  Participants will be queried regarding their analgesic use over the past week (for all participants including those prescribed an opioid/other analgesic from non-study providers) to determine morphine equivalents. Adherence to prescription medication instructions will be monitored by self-report. This outcome will be applicable to: Phase 1- participants prescribed opioids prior to study initiation; Phase 2- participants prescribed opioids prior to study initiation and those who receive an opioid prescription from a study clinician during the course of the study or longer-term follow-up.
Time to receipt of additional treatment for to KOA | Up to 2 years
  Healthcare utilization will be measured as it relates to KOA on an ongoing basis throughout the study
Treatment response as a binary outcome for Phase 1 and 2 intervention arms using the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) guidelines | Opioid use and pain are measured at all follow-up time points and will be used through Phase1: 8 weeks post-rand. and 8 weeks post-treatment; Phase 2: 12 weeks post-rand. and 8 weeks post-treatment
  BPI intensity will be measured, per IMMPACT cut off guidelines and will also incorporate changes in opioid dose. A 20% decrease in pain intensity is minimally important, ⩾30% moderately important and ⩾50% substantial. Each of these brackets will be evaluated to determine responders at the pain criteria cut points.
  Despite meeting guideline criteria, anyone meeting the following will not be considered a treatment responder:
  1. Increase in new opioid use of >15 morphine milligram equivalents (MME) or;
  2. Increase of >100mg Tramadol
Treatment response as a binary outcome for Phase 1 and 2 intervention arms based on OARSI-OMERACT guidelines, incorporating changes in opioid dose. | Opioid use and pain assessed up to 2 years. PGIC assessed at main outcome visit (8 and 12 weeks for Phase 1 and Phase 2, respectively). The treatment response categorical outcome will be analyzed separately for mITT and per- protocol analyses.
  BPI intensity, KOOS, PGIC and opioid use will be measured, and define a categorical outcome based on Osteoarthritis Research Society International (OARSI) Standing Committee for Clinical Trials Response Criteria Initiative and the Outcome Measures in Rheumatology (OARSI-OMERACT) guidelines (pain, function measures, and patient assessment), incorporating changes in opioid dose.
  A treatment responder will be defined as either:
  High improvement in pain or in function ≥50% and absolute change of >2 for BPI and ≥20 for KOOS,
  Or
  Improvement in at least 2 of the 3 following:
  * pain ≥20% and absolute change of >1
  * function ≥20% and absolute change ≥10
  * patient's global impression of change ≥minimal improvement
  Despite meeting guideline criteria, anyone meeting the following will not be considered a treatment responder:
  1. Increase in new opioid use of >15 morphine milligram equivalents (MME) or;
  2. Increase of >100mg Tramadol

CONTACTS AND LOCATIONS:
Overall Officials: Steven Cohen, MD, Principal Investigator — Johns Hopkins University
Locations (24):
- United States (24):
  - University of California Davis, Sacramento, California
  - University of California San Diego, San Diego, California
  - VA Medical Center San Diego, San Diego, California
  - University of Colorado, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins, Baltimore, Maryland
  - Walter Reed Army Medical Center, Bethesda, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Weill Cornell University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Cleveland VA Medical Center, Cleveland, Ohio
  - University Hospitals, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Vanderbilt University, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Upon completing data collection, specifically after the last patient's main outcome visit (excluding long-term follow-up), the HEAL Pain Management Effectiveness Research Network (ERN) Data Coordinating Center (DCC) at the University of Utah will compile the final study dataset. This dataset will undergo statistical analyses and form the basis for publishing both primary and secondary trial results. The SKOAP dataset, recognized as valuable for pain management and opioid use research communities, will be formatted for accessibility to non-ERN investigators. Additionally, a data dictionary will accompany the dataset, offering concise definitions for each included data element. Any peculiarities impacting interpretation or analysis will be outlined within the dictionary. Unreliable data elements will be removed, with documentation provided accordingly.
Supporting Information: Study Protocol
Time Frame: These policies are expected to focus primarily on the timing of data release. The investigators preliminary plan is to release the database (defined below) and supporting information at the time of publication of the primary manuscript, or within 12 months of last patient's final follow-up, whichever comes first. Implementation of the plan will follow the HEAL Public Access and Data Sharing Policy as outlined at https://heal.nih.gov/about/public-access-data.
Access Criteria: Access to the releasable database housed in the NIH-assigned repository will be in accordance with procedures and regulations of the NIH or specific institute. The data coordinating center will not provide any support for investigators using the releasable database.

DOCUMENTS (1):
  • Informed Consent Form (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/12/NCT04504812/ICF_000.pdf